CLINICAL TRIAL: NCT01932138
Title: Evaluation of Interventions to Achieve Universal Access to PMTCT Services and Reduce Mother-to-Child Transmission of HIV in Dar es Salaam, Tanzania
Brief Title: Trial to Improve Access to PMTCT Services and Reduce HIV Transmission From Mother to Child
Acronym: FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Management and Development for Health, Tanzania (Unknown); Elton John AIDS Foundation (Other); Comic Relief UK (Unknown)
Responsible Party: Principal Investigator, Till Barnighausen, Associate Professor of Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EJF22802
Record Dates: First submitted 2013-05-14; First posted 2013-08-30 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Mother-to-child Transmission of HIV; Pregnancy
Keywords: Community-based intervention; Community health workers; Antenatal care; HIV; PMTCT; HIV vertical transmission; Public-sector health systems
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced CHW intervention (Experimental): CHWs will 1) identify pregnant women through home visits and refer them to ANC; 2) inform pregnant women on antenatal care ANC and PMTCT; 3) visit women at home to ascertain ANC attendance; and 4) follow up women who have missed ANC or PMTCT appointments.
  Interventions: Other: Enhanced CHW intervention
- Standard of care (Other): Clinic-based health workers follow-up patients who have missed scheduled PMTCT appointments (through telephone calls and/or in-person visits). The standard of care does not include any specific interventions to improve ANC attendance.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Enhanced CHW intervention — The CHW employed in this study are a health worker cadre that already exists in the Tanzanian public-sector health system, so-called "home-base carers" (or HBC). The HBC in this study are supervised by another existing cadre, so-called "community-based health care workers" (or CBHC). The CBHC are clinic-based and are charged to organize community outreach activities in the Tanzanian public-sector health systems. The CBHC (1-2 per clinic) are also active in the control arm; in this intervention arm, there role is changed: they are actively supervising a large number of CHW. Per street (or mtaa), 1-2 CHW are assigned to carry out the enhanced CHW intervention.
  Arms: Enhanced CHW intervention
Other: Standard of care — The standard of care in the Tanzanian health care system does not include any CHW intervention to enhance ANC and PMTCT uptake and retention. The only community-based intervention are PMTCT follow-up organized by a health worker cadre who works out of ANC and primary care clinics (so-called CBHC).
  Arms: Standard of care

SUMMARY:
The purpose of this study is to determine the effectiveness, cost-effectiveness, feasibility and acceptability of an enhanced community health worker (CHW) intervention and outreach system to improve antenatal care and PMTCT uptake and retention, and to decrease mother-to-child HIV transmission.

DETAILED DESCRIPTION:
Mother-to-child transmission of HIV/AIDS (MTCT) is still a major contributor to the burden of HIV infections among infants and children in Sub-Saharan Africa. Among the major challenges of each approach to achieving maximum benefits is late and incomplete antenatal care (ANC) attendance. While attendance to one ANC visit is almost universal, only about half of pregnant women attend the four WHO-recommended visits. Moreover, those that attend often book late in pregnancy. This nationwide challenge can lead to delays or interferences with the appropriate PMTCT medications for mothers -thus substantially diminishing the potential of PMTCT care to reduce mother-to child-transmission of HIV in Tanzania.

The investigators will examine the effectiveness, cost-effectiveness, feasibility, and acceptability of an enhanced community health worker intervention and outreach system for pregnant women to facilitate early and consistent ANC attendance, early and effective PMTCT uptake, with the aim to further reduce mother-to-child transmission of HIV. We will test the effectiveness hypothesis in a cluster-randomized controlled trial; the unit of randomization is the administrative unit of a ward, which is the geographical unit below a district in the Tanzanian government system. We randomly allocate all 60 wards in two of the three districts in Dar es Salaam, Tanzania -- Kinondoni and Ilala districts -- to receiving the enhanced community health worker intervention and outreach system vs. receiving the standard of care in the Tanzanian public-sector health system.

The results of this study will inform implementers and policy makers on whether and how a community outreach system and PMTCT algorithm may maximize benefits of antenatal care and PMTCT services in Tanzania and inform decisions surrounding future maternal and newborn health programs moving forward.

This study was initially designed to test both the effectiveness of the enhanced CHW intervention and outreach system and the effectiveness of WHO PMTCT option B (vs. A) in ensuring successful PMTCT in the Tanzanian public-sector health system. However, in reaction to a report of non-compliance by the investigator team (incomplete records of written informed consent among PMTCT patients in the public-sector PMTCT clinics) the IRB at the Harvard School of Public Health decided to stop involvement in the option A vs. B component of this study. The IRB approved continuation of the enhanced CHW intervention and outreach system in the study.

ELIGIBILITY:
Inclusion Criteria:

• All pregnant women who are identified by the CHW during the routine household visits

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190530 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of infants born to HIV-infected mothers who have acquired HIV | During the first 2 years of life
Proportion of HIV-exposed infants tested for HIV | During the first 2 years of life
Proportion of pregnant women making at least four antenatal clinic visits | Between the first week of gestation and delivery
Proportion of pregnant women delivering at a healthcare facility | At delivery
Proportion of HIV-positive women receiving PMTCT | Between the first antenatal care visit and 1 week after stopping breastfeeding

SECONDARY OUTCOMES:
Number of weeks of gestation at which pregnant women have their first ANC visit | Between the first week of gestation and delivery
Proportion of HIV-infected pregnant women who completed PMTCT | Between the first antenatal care visit and 1 week after stopping breastfeeding
Proportion of HIV-exposed infants who received PMTCT | During the first 2 years of life
Proportion of pregnant women who were tested for HIV | Between the first week of gestation and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, MD ScD, Principal Investigator — Harvard School of Public Health (HSPH); Guerino Chalamilla, MD PhD, Principal Investigator — Management and Development for Health
Locations (1):
- Management and Development for Health, Dar es Salaam, Tanzania

REFERENCES:
- [Background] Sando D, Geldsetzer P, Magesa L, Lema IA, Machumi L, Mwanyika-Sando M, Li N, Spiegelman D, Mungure E, Siril H, Mujinja P, Naburi H, Chalamilla G, Kilewo C, Ekstrom AM, Fawzi WW, Barnighausen TW. Evaluation of a community health worker intervention and the World Health Organization's Option B versus Option A to improve antenatal care and PMTCT outcomes in Dar es Salaam, Tanzania: study protocol for a cluster-randomized controlled health systems implementation trial. Trials. 2014 Sep 15;15:359. doi: 10.1186/1745-6215-15-359. PMID 25224756
- [Derived] Geldsetzer P, Mboggo E, Larson E, Lema IA, Magesa L, Machumi L, Ulenga N, Sando D, Mwanyika-Sando M, Spiegelman D, Mungure E, Li N, Siril H, Mujinja P, Naburi H, Chalamilla G, Kilewo C, Ekstrom AM, Foster D, Fawzi W, Barnighausen T. Community health workers to improve uptake of maternal healthcare services: A cluster-randomized pragmatic trial in Dar es Salaam, Tanzania. PLoS Med. 2019 Mar 29;16(3):e1002768. doi: 10.1371/journal.pmed.1002768. eCollection 2019 Mar. PMID 30925181